CLINICAL TRIAL: NCT05731141
Title: A Prospective Natural History Study of Lymphatic Anomalies
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001084; 001084-CH
Record Dates: First submitted 2023-02-15; First posted 2023-02-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11-26

CONDITIONS: Lymphatic Diseases; Lymphatic Abnormalities
Keywords: Protein Losing Enteropathy; Lymphedema; Lymphangiectasia; Kaposiform Lymphangiomatosis; Gorham Stout Disease; Generalized Lymphatic Anomaly; Complex Lymphatic Anomaly; Chylous Effusion; Chylous Ascites; Central Conducting Lymphatic Anomaly
MeSH Terms: conditions — Lymphatic Diseases; Lymphatic Abnormalities; Protein-Losing Enteropathies; Lymphedema; Lymphangiectasis; Osteolysis, Essential; Chylous Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Degree Relatives: Siblings or parents of patients.
- Patients: Patients with lymphatic anomalies.

SUMMARY:
Background:

The lymphatic system is a network of vessels that carry a clear fluid called lymph through the body. Problems in the lymphatic system can cause pain, fluid buildup, and issues with immunity. There is much researchers do not understand about lymphatic anomalies. In this natural history study, they will collect data from a lot of people over a long time.

Objective:

To better understand why lymphatic anomalies develop. The goal is to improve future treatments.

Eligibility:

People aged 0 days and older with a suspected or confirmed lymphatic anomaly. Their unaffected parents or siblings aged 7 years or older are also needed.

Design:

Participants may remain in the study indefinitely. Affected participants may be evaluated every 10 months to 2 years. Some participants will be seen over telemedicine. Others will be seen at the NIH Clinical Center for 2-5 days.

All participants will have a physical exam. They may provide specimens including blood, saliva, hair follicles, stool, skin, and other tissues. Samples may be used for genetic testing.

Participants may undergo other tests depending on their medical conditions. The NIH Clinical Center visit may include:

Heart tests include placing stickers on the chest to measure electrical activity and using sound waves to capture pictures of the heart.

A lung test measures the muscle strength in the chest. Participants will blow into a tube.

Photographs may be taken of participants faces and other features.

Imaging scans will take pictures of the inside of the body. One scan will measure bone density.

One type of scan tracks how lymph fluid moves through the body. Participants will be under anesthesia, and they will be injected with a dye.

DETAILED DESCRIPTION:
Study Description:

A natural history study for lymphatic anomalies to systematically evaluate the disease phenotypes and long-term outcomes to provide improved prognostication to families, establish screening/monitoring guidelines, determine best practices for genetic diagnosis, explore family opinions, and explore fertility for those on long term medication management. This study will allow us to identify novel end points for future clinical trials.

Objectives:

Primary objectives:

* To establish a longitudinal cohort of participants with lymphatic anomalies
* To longitudinally determine the age at presentation and incidence of clinical features

Secondary objectives:

* To establish a longitudinal biospecimen repository
* To determine the best practices for genetic diagnosis based on phenotype.
* To determine the malignant potential of anomalies longitudinally

Endpoints:

Primary endpoints:

* The number of participants with lymphatic anomalies
* For each clinical feature or symptoms, the range of ages at the development of that feature/symptom and fraction of participants with that feature
* Quantification and identification of novel features associated with disease.

Secondary endpoints:

* The number of specimens collected
* Diagnostic yields by phenotype and genetic test methodology
* Number of malignancies related to the primary lesion that have developed

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected (Proband)

In order to be eligible to participate in this study, an individual must meet one of the following criteria as determined after review of medical history:

* Current or history of lymphatic anomaly or symptoms suggestive of a lymphatic disorder Or
* An ill-defined vascular anomaly that is suspected to have an abnormal lymphatic component Or
* A pathogenic, likely pathogenic, or VUS in a genetic disorder with a known lymphatic component Or
* Clinical diagnosis of a syndrome with a known lymphatic component

Unaffected (First Degree Relatives: Parents and Siblings)

Genetic variants underlying complex lymphatic anomalies can be passed down through parents or be new in a child (de novo). Inclusion of first-degree relatives will assist in genetic analysis to delineate whether the variant is inherited or de novo.

To be eligible to participate as a first degree relative in this study, an individual must be a first-degree family member of an affected participants

EXCLUSION CRITERIA:

Affected Proband

An individual who meets any of the following criteria will be excluded from participation in this study after review of medical history, concomitant medication and allergy review, anthropometrics, and performance status:

-Any condition, in the opinion of the investigator, that would increase risk of participation or impair their ability to comply with protocol requirements.

Lymphatic anomalies that are definitively determined to be secondary by the principal investigator will be excluded from this study. For example, participants who develop a lymphedema after breast cancer surgery.

Unaffected (First Degree Relatives)

-Any condition, in the opinion of the investigator, that would increase risk of participation or impair their ability to comply with protocol requirements.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lymphatic anomalies and their parents.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish a longitudinal cohort of participants with lymphatic anomalies | 12/31/2028
  We plan to enroll a group of participants willing to participate in the study over time.
To longitudinally determine the age at presentation and incidence of clinical features | 12/31/2028
  For each clinical feature or symptoms, the range of ages at the development of that feature/symptom and fraction of participants with that feature

SECONDARY OUTCOMES:
To establish a longitudinal biospecimen repository | 12/31/2028
  We plan to collect biospecimens including, but not limited to blood and stool from participants over time.
To determine the best practices for genetic diagnosis based on phenotype | 12/31/2028
  We will analyze diagnostic yields by phenotype (how many participants are able to have a genetic diagnosis in proportion to the number of participants who receive genetic testing) and genetic test methodology (to determine which genetic test is most helpful in diagnosing lymphatic anomalies)
To determine the malignant potential of anomalies longitudinally | 12/31/2028
  We will track the number of malignancies related to the primary lesion that have developed

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Sheppard, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share human data generated in this research for future research as follows:@@@@@@De-identified data in an NIH-funded or approved public repository. @@@@@@De-identified data in another public repository. @@@@@@De-identified data in BTRIS (automatic for activities in the Clinical Center)@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.
Supporting Information: CSR
Time Frame: At the time of publication or shortly thereafter.
Access Criteria: Data will be shared through:@@@@@@An NIH-funded or approved public repository: clinicaltrials.gov @@@@@@BTRIS (automatic for activities in the Clinical Center)@@@@@@Approved outside collaborators under appropriate individual agreements.@@@@@@Publication and/or public presentations.@@@@@@This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers after the completion of the primary endpoint by contacting Sarah Sheppard, PI of the study.

REFERENCES:
- [Background] Makinen T, Boon LM, Vikkula M, Alitalo K. Lymphatic Malformations: Genetics, Mechanisms and Therapeutic Strategies. Circ Res. 2021 Jun 25;129(1):136-154. doi: 10.1161/CIRCRESAHA.121.318142. Epub 2021 Jun 24. PMID 34166072
- [Background] Brouillard P, Witte MH, Erickson RP, Damstra RJ, Becker C, Quere I, Vikkula M. Primary lymphoedema. Nat Rev Dis Primers. 2021 Oct 21;7(1):77. doi: 10.1038/s41572-021-00309-7. PMID 34675250
- [Background] Liu M, Smith CL, Biko DM, Li D, Pinto E, O'Connor N, Skraban C, Zackai EH, Hakonarson H, Dori Y, Sheppard SE. Genetics etiologies and genotype phenotype correlations in a cohort of individuals with central conducting lymphatic anomaly. Eur J Hum Genet. 2022 Sep;30(9):1022-1028. doi: 10.1038/s41431-022-01123-9. Epub 2022 May 24. PMID 35606495
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001084-CH.html